CLINICAL TRIAL: NCT03389893
Title: Effect of Dupilumab (Anti-IL4Rα) on the Host-Microbe Interface in Atopic Dermatitis, Dupilumab Study
Brief Title: Effect of Dupilumab (Anti-IL4Rα) on the Host-Microbe Interface in Atopic Dermatitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to inability to meet accrual goals within the funding period.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Regeneron Pharmaceuticals (Industry); Sanofi (Industry); Atopic Dermatitis Research Network (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ADRN-09; U19AI117673 (NIH); NIAID DAIT CRMS ID#: 38439 (Other: DAIT NIAID)
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis (AD)
Keywords: randomized double-masked (blind) placebo-controlled trial; T helper 2 (Th2) effect; cutaneous microbial community; skin barrier
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab w/OLE (Experimental): Participants will receive a loading dose of dupilumab (two 300 mg subcutaneous (subcut) injections (total of 600 mgs)) on Day 0, followed by 300 mg dose of dupilumab by subcut injection every 2 weeks (Days 14 and 28).
  Open Label Extension (OLE): Participants will begin a 10 week OLE on Day 42, beginning with a loading dose of two subcut administered injections (one 300 mg dose of dupilumab and one dose of placebo, in order to protect prior masking/blind).Participants will then maintain a regimen of 300 mg of dupilumab by subcut injection every two weeks through Day 98.
  The subcut injections will be administered in the abdomen (except for the 2 inches (5 cm) around the navel-not allowed), thighs, or upper arms. Injection sites will be rotated with each dose.
  Interventions: Drug: Dupilumab; Drug: Placebo
- Placebo Comparator w/OLE (Placebo Comparator): Participants will receive a loading dose of placebo (two placebo subcutaneous (subcut) injections) on Day 0 followed by one dose of placebo by subcut injections every 2 weeks (Days 14 and 28).
  Open Label Extension (OLE): Participants will begin a 10 week OLE on Day 42, beginning with a loading dose of dupilumab (two 300 mg subcut injections (total of 600 mgs)-protection of prior masking/blind maintained). Participants will then maintain a regimen of 300 mg of dupilumab by subcut injection every two weeks through Day 98.
  The subcut injections will be administered in the abdomen (except for the 2 inches (5 cm) around the navel-not allowed), thighs, or upper arms. Injection sites will be rotated with each dose.
  Interventions: Drug: Dupilumab; Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Dupilumab, an interleukin (IL)-4 receptor alpha (IL-4Rα) antagonist, is indicated for the treatment of adult patients with moderate-to-severe atopic dermatitis whose disease is not adequately controlled with topical prescription therapies or when those therapies are not advisable. (FDA approved on March 28, 2017.)
  Other Names: Dupixent®; IL4Ra mAb
Drug: Placebo — Placebo will contain the identical formulation as the dupilumab formulation without the active mAb and will be given by exactly the same route and schedule through Day 28.
  Other Names: Dupilumab placebo

SUMMARY:
The purpose of this study is to understand the effect that T helper 2 (Th2) blockade has on well-described pathophysiological features of Atopic Dermatitis (AD), for example: barrier, epidermal activation, dysbiosis and epidermal lipids.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-masked, placebo-controlled trial investigating the effect of 6 weeks of dupilumab treatment on quantitative and qualitative measures of cutaneous microbial community structure, skin barrier biology, and circulating T cell profiles, in adults with chronic moderate-to-severe atopic dermatitis (AD).

After obtaining informed consent, eligible participants will return to clinic for their Treatment Initiation Visit (Day 0) and will be randomized 2:1 active to placebo. Participants will receive three doses of dupilumab or placebo based on their randomization assignment. The first dose (600 mg loading dose of dupilumab or placebo) will be administered on Day 0 and the second and third doses (300 mg dupilumab or placebo) on Day 14 and Day 28, respectively.

Participants will return to clinic on Days 3, 7, and 21 during the double-masked portion of the study. Participants will begin the open-label extension (OLE) at Day 42 and will receive dupilumab (600 mg loading dose [two 300 mg injections] for those initially randomized to the placebo group and a 300 mg dose plus placebo injection for those initially randomized to the dupilumab group). Participants will return to clinic on Days 77 and 112 during the OLE portion of the study. During all visits (Day 0-Day 112), Adverse Events (AEs), concomitant medications, and medical history will be assessed and physical exams including assessment of AD severity will be performed. Blood, urine, skin swabs, skin tape strips, and skin biopsies, as applicable, will be collected, and barrier assessments will be performed per the Schedule of Events, per protocol. Samples will be collected prior to dupilumab or placebo administration on Days 0, 14, 28, and 42. After Day 112, a follow-up call (Day 182) will be made to assess for pregnancy, current medications, and adverse events (AEs).

If concerns arise between regularly scheduled visits, participants will be instructed to contact study personnel and may be asked to return to the study site for an "Unscheduled Visit." Participants may be asked to return for Unscheduled Visits, as needed for the duration of the study, to provide additional blood, skin swabs, skin tape strips, or skin biopsies,as applicable, for further mechanistic and functional studies, if biosamples are lost or destroyed, or if insufficient yields were obtained at a previous study visit.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and provide informed consent
* Chronic AD, (according to the Atopic Dermatitis Research Network [ADRN] Standard Diagnostic Criteria), that has been present for at least 3 years before the Screening Visit
* EASI score ≥12 at the Screening Visit and ≥16 at the Treatment Initiation Visit
* Investigator Global Assessment (IGA) score ≥3 (on the 0-4 IGA scale) at the Screening and Treatment Initiation Visits
* ≥10% body surface area of AD involvement at the Screening and Treatment Initiation Visits
* Must have active lesions (minimum of 3 of at least 4x4 cm^2 each on the upper or lower extremities, excluding the palms of the hands and soles of the feet) at the Screening and Treatment Initiation Visits
* Documented recent history (within 6 months before the Screening Visit) of inadequate response to outpatient treatment with topical corticosteroids of medium to high potency (± topical calcineurin inhibitors as appropriate), or for whom topical treatments are otherwise inadvisable
* Must agree to apply a stable dose of a topical emollient (moisturizer) at least twice daily for at least 7 days before the Treatment Initiation Visit, and must confirm application at the Treatment Initiation Visit
* Individuals with asthma must adhere to asthma controller medication(s) for the duration of the study including the open-label and follow-up portions
* Females of childbearing potential must have a negative pregnancy test at the Screening and Treatment Initiation Visits
* Females with reproductive potential* and sexually active must agree to use FDA approved methods of birth control for the duration of the study, including during the open-label and follow-up portions of the study:

  --FDA approved methods of birth control include hormonal contraceptives, intrauterine device, double barrier contraception (i.e., condom plus diaphragm), or male partner with documented vasectomy.

  ---*Menopause is defined as at least 12 consecutive months without menses; if in question, a follicle stimulating hormone of ≥25 U/mL must be documented. Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable; if documented, women with these conditions are not required to use additional contraception.
* Males who are sexually active must agree to use an acceptable method of birth control (e.g. barrier methods with vaginal spermicide, surgical sterilization or surgically sterilized partner), or have a female partner practicing an approved birth control method for females as described in Inclusion Criterion above.
* Willing and able to comply with all clinic visits and study-related procedures
* Able to understand and complete study-related questionnaires

Exclusion Criteria:

* Inability or unwillingness of an individual to give written informed consent or comply with study protocol
* Known systemic hypersensitivity to any of the excipients of the dupilumab or placebo study products
* Known or suspected immunosuppression, including history of invasive opportunistic infections (e.g., tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution, or otherwise recurrent immune-compromised status, as judged by the investigator
* Known history of human immunodeficiency virus (HIV) infection
* Ocular disorder that, in the opinion of the investigator, could adversely affect the individual's risk for study participation. Examples include, but are not limited to, individuals with a history of or active case of:

  * herpes keratitis,
  * Sjogren's Syndrome,
  * keratoconjunctivitis sicca or Dry Eye Syndrome that requires daily use of supplemental lubrication, or
  * ocular condition(s) requiring the regular use of ocular corticosteroids or cyclosporine.
* Parasitic infection, except for vaginal trichomoniasis, within 12 months of the Treatment Initiation Visit, or high risk for contracting parasitic infections (e.g., living in or traveling to endemic areas)
* Presence of skin comorbidities that may interfere with study assessments
* History of malignancy within 5 years before the Treatment Initiation Visit except completely treated in situ carcinoma of the cervix, and completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin or melanoma in situ
* History of non-malignant lymphoproliferative disorders
* History of alcohol or drug abuse within 2 years before the Screening Visit
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the individual's participation in the study. Examples include, but are not limited to, individuals with short life expectancy, uncontrolled diabetes (HbA1c ≥9%), cardiovascular conditions (e.g., stage III or IV cardiac failure according to the New York Heart Association classification), severe renal conditions (e.g., individuals on dialysis), hepato-biliary conditions (e.g., Child-Pugh class B or C), neurological conditions (e.g., demyelinating diseases), active major autoimmune diseases (e.g., lupus, inflammatory bowel disease, rheumatoid arthritis, etc.), other severe endocrinological, gastrointestinal, metabolic, pulmonary, or lymphatic diseases.
* Any other medical or psychological condition including relevant laboratory abnormalities at screening that, in the opinion of the investigator, suggests a new and/or insufficiently understood disease, may present an unreasonable risk to the study participant as a result of his/her participation in this clinical trial, may make individual's participation unreliable, or may interfere with study assessments. This includes hypersensitivity to local anesthetics (e.g., lidocaine or Novocain), bleeding disorders, treatment with anticoagulants or other conditions that make the biopsy procedure inadvisable.
* Planned major surgical procedure during the screening period or study treatment (i.e. Screening through Day 112)
* Member of the investigational team or his/her immediate family
* Pregnant or breast-feeding women, or women planning to become pregnant or breastfeed during the study including the open-label and follow up portions of the study
* Individuals unwilling to use adequate birth control, if of reproductive potential and sexually active. Adequate birth control is defined as agreement to consistently practice an approved method of contraception for the duration of the study, including the open-label and follow up portions of the study.
* History of keloid formation
* History of serious life-threatening reaction to latex, tape, or adhesives
* Prior treatment with dupilumab
* Individuals with asthma who have required use of a systemic corticosteroid within 3 months prior to the Treatment Initiation Visit or who require a dose greater than 880 mcg/day of fluticasone propionate or equivalent inhaled corticosteroid to maintain asthma control
* Treatment with biologics as follows:

  * Any cell-depleting agents, including but not limited to rituximab, within 6 months before the Treatment Initiation Visit, or until lymphocyte and CD 19+ lymphocyte count returns to normal, whichever is longer
  * Infliximab, adalimumab, golimumab, certolizumab pegol, abatacept, etanercept, anakinra within 16 weeks before the Treatment Initiation Visit for any indication, or
  * Other biologics within 5 half-lives (if known) or 16 weeks before the Treatment Initiation Visit, whichever is longer
* Treatment with a live (attenuated) vaccine within 12 weeks before the Treatment Initiation Visit or planning to receive a live vaccine during the study (through Day 182)
* Use of an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the Treatment Initiation Visit
* Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks before the Treatment Initiation Visit, or superficial skin infections within 1 week before the Treatment Initiation Visit
* The following treatments within 4 weeks before the Treatment Initiation Visit, or any condition that, in the opinion of the investigator, will likely require such treatment(s) during the screening period and study treatment (i.e., Screening through Day 112):

  * Systemic corticosteroids
  * Immunosuppressive/immunomodulating drugs (e.g., cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, or methotrexate)
* Use of phototherapy (such as narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + UVA [PUVA]) or a tanning booth/parlor within 4 weeks of the Treatment Initiation Visit
* Treatment with bleach bath within 3 weeks before the Treatment Initiation Visit
* Use of a chlorinated hot tub within 3 weeks before the Treatment Initiation Visit
* Treatment with topical corticosteroids, phosphodiesterase inhibitors (crisaborole), or calcineurin inhibitors (tacrolimus or pimecrolimus) within 1 week before the Treatment Initiation Visit
* Initiation of treatment of AD with prescription moisturizers or moisturizers containing ceramide, hyaluronic acid, urea, or filaggrin during the screening period (participants may continue using stable doses of such moisturizers if initiated before the Screening Visit)
* Planned or anticipated use of any prohibited medications or procedures during the screening period and study treatment (i.e., Screening through Day 112)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Beck, MD, Study Chair — University of Rochester
Locations (9):
- United States (9):
  - University of California San Diego, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Rochester Medical Center, Rochester, New York
  - Duke University, Durham, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- See also: National Institute of Allergy and Infectious Disease (NIAID) Website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 participants were randomized from July 2018 to March 2020 from 9 clinical sites.First participant enrollment occurred on July 25, 2018.
Pre-assignment Details: Informed consent was obtained from potentially eligible individuals who underwent a screening visit to determine eligibility.
Groups:
- Dupilumab: Participants received a loading dose of two 300 mg subcutaneous injections on Day 0 followed by 300 mg subcutaneous injections every two weeks (Days 14 and 28).
- Placebo: Placebo contained the identical formulation as the dupilumab formulation without the active monoclonal antibody and was given by exactly the same route and schedule through Day 28.
- Dupilumab to Open-Label Extension Dupilumab: Open Label Extension (OLE): Participants started a 10 week OLE on Day 42, beginning with a loading dose of two subcutaneously administered injections (one 300 mg dose of dupilumab and one dose of placebo, in order to protect prior masking/blind). Participants then maintained a regimen of 300 mg of dupilumab by subcutaneous injection every two weeks through Day 98. The participants then entered a follow-up period until Day 182.
- Placebo to Open-Label Extension Dupilumab: Open Label Extension (OLE): Participants started a 10 week OLE on Day 42, beginning with a loading dose of dupilumab (two 300 mg subcutaneous injections [total of 600 mg]-protection of prior masking/blind maintained). Participants then maintained a regimen of 300 mg of dupilumab by subcutaneous injection every two weeks through Day 98. The participants then entered a follow-up period until Day 182.
Period: Randomized Double Blind Period
Arm/Group | Dupilumab | Placebo | Dupilumab to Open-Label Extension Dupilumab | Placebo to Open-Label Extension Dupilumab
Started (The primary outcome was measured through Day 28, during the Randomized Double Blind Placebo Controlled (RDBPC) portion of the study.) | 46 | 26 | 0 | 0
Completed | 45 | 26 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Open Label Extension and Follow-Up
Arm/Group | Dupilumab | Placebo | Dupilumab to Open-Label Extension Dupilumab | Placebo to Open-Label Extension Dupilumab
Started | 0 | 0 | 45 | 26
Completed (3 participants were lost to follow-up after Day 112) | 0 | 0 | 41 | 25
Not Completed | 0 | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Participant Moved | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT): All participants who were randomized and have Staphylococcus aureus (S. aureus) abundance measured at Day 0 and Day 28.
Groups:
- Dupilumab+Open Label Extension and Follow-Up: Participants received a loading dose of two 300 mg subcutaneous injections on Day 0 followed by 300 mg subcutaneous injections every two weeks (Days 14 and 28). Participants started a 10 week OLE on Day 42, beginning with a loading dose of two subcutaneously administered injections (one 300 mg dose of dupilumab and one dose of placebo, in order to protect prior masking/blind). Participants then maintained a regimen of 300 mg of dupilumab by subcutaneous injection every two weeks through Day 98. The participants then entered a follow-up period until Day 182.
- Placebo+Open Label Extension and Follow-Up: Placebo contained the identical formulation as the dupilumab formulation without the active monoclonal antibody and was given by exactly the same route and schedule through Day 28. Participants started a 10 week OLE on Day 42, beginning with a loading dose of dupilumab (two 300 mg subcutaneous injections [total of 600 mg]-protection of prior masking/blind maintained). Participants then maintained a regimen of 300 mg of dupilumab by subcutaneous injection every two weeks through Day 98. The participants then entered a follow-up period until Day 182.
- Total: Total of all reporting groups
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up | Total
Number analyzed (Participants) | 45 | 26 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (15.56) | 37.3 (15.61) | 36.8 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 7 | 24
  Male | 28 | 19 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 39 | 22 | 61
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 21 | 13 | 34
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 26 | 71
Body Weight [Mean (Standard Deviation); unit: kilograms (Kg)] — Participant weight measured at the Screening Visit.
  kilograms (Kg) | 80.7 (19.45) | 79.4 (18.58) | 80.2 (19.01)
Height [Mean (Standard Deviation); unit: centimeters (Cm)] — Participant height measured at the Screening Visit.
  centimeters (Cm) | 170.9 (9.27) | 175.3 (11.74) | 172.5 (10.38)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Participant BMI measured at the Screening Visit.
  Kg/m^2 | 27.5 (5.69) | 25.7 (4.90) | 26.9 (5.45)
SCORing Atopic Dermatitis (SCORAD) [Mean (Standard Deviation); unit: units on a scale] — SCORAD is a composite severity index comprising a) the amount/extent of body surface area affected, b) subjective symptom visual analog assessments of itch and sleep loss [itch: 0 = no itch to 10 = worst itch imaginable and sleep loss: 0=no sleep loss to 10=worst imaginable sleep loss], and c) 6 disease intensity assessments [dryness, erythema, edema/papulation, excoriation, lichenification and oozing/crusting] each graded from 0-3: 0=none, 1=mild, 2=moderate and 3=severe. SCORAD is scored from 0=no AD present to 103=severe. The reported value is from the treatment initiation visit (Day 0).
  units on a scale | 62.1 (11.7) | 59.9 (10.86) | 61.3 (11.38)
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — EASI is a composite score (range:0-72) measuring physical signs of atopic dermatitis,including area of involvement and severity.Severity components include: erythema, papulation, excoriation and lichenification [0=absent, 1=mild, 2=moderate, 3=severe] for each body region (head/neck, trunk, arms, legs). Area of involvement (%) is assessed for each body region. Area and severity of each body region is weighted based on size of region, and region scores are added for the total score[≤7=mild, >7 and ≤21.1=moderate, >21.1=severe].The reported value is from the treatment initiation visit (Day 0).
  units on a scale | 28.4 (12.16) | 28.6 (10.89) | 28.5 (11.63)
Eczema Area and Severity Index (EASI) Score < 21.1 [Count of Participants; unit: Participants] — Dichotomous variable based on EASI score (range:0-72) used as a stratification factor during randomization to differentiate severe (>21) and non-severe (≤21). The reported value is from the treatment initiation visit (Day 0).
  Participants | 16 | 10 | 26
Nottingham Eczema Severity Score [Mean (Standard Deviation); unit: units on a scale] — The Nottingham Eczema Severity Score assesses the clinical severity of atopic dermatitis base on the clinical duration, intensity as measured by sleep disturbance, and the extent of disease involvement. Each parameter is scored from 1-5, and the individual scores are added to obtain the total score. Scores between 3 and 8 are considered mild, between 9 and 11 are considered moderate, and between 12 and 15 are considered severe. The reported value is from the treatment initiation visit (Day 0).
  units on a scale | 13.5 (1.49) | 13.6 (1.21) | 13.5 (1.38)
Investigator Global Assessment (IGA) [Count of Participants; unit: Participants] — Investigator Global Assessment (IGA) score is a subjective scale measuring disease severity. Based on a 5-point scale from 0 (completely clear) to 4 (severe). Defined score of 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe. The reported value is from the treatment initiation visit (Day 0).
  Participants
    Moderate | 16 | 11 | 27
    Severe | 29 | 15 | 44
Average itch in the past 24 hours as assessed by Pruritus Numerical Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Pruritus NRS scale is an assessment tool that is used to report the average intensity of a participant's pruritus (itch) during a 24-hour recall period. Participants were asked to report the average itch experienced during the past 24 hours on a scale of 0 - 10 [0= no itch; 10= worst imaginable itch]). The reported value is from the treatment initiation visit (Day 0).
  units on a scale | 6.7 (2.17) | 7.0 (1.48) | 6.8 (1.94)
Self-reported history of Eczema Herpeticum [Count of Participants; unit: Participants] — Participants were asked the following question at the screening visit: 'Have you ever been diagnosed with Eczema Herpeticum by a health care provider?' Participants who responded 'yes' were counted.
  Participants | 1 | 1 | 2
Self-reported history of Staph infection [Count of Participants; unit: Participants] — Participants were asked the following question at the screening visit: 'Have you ever had a Staph infection?' Participants who responded 'yes' were counted.
  Participants | 15 | 9 | 24
Self-reported history of food allergy [Count of Participants; unit: Participants] — Participants were asked the following question at the treatment initiation visit (Day 0): 'Do you have known past or current history of food allergies?' Participants who responded 'yes' were counted.
  Participants | 15 | 14 | 29
Self-reported history of animal allergies [Count of Participants; unit: Participants] — Participants were asked the following question at the treatment initiation visit (Day 0): 'Do you have known allergies to animals?' Participants who responded 'yes' were counted.
  Participants | 30 | 19 | 49
Self-reported pets living in the participant's home [Count of Participants; unit: Participants] — Participants were asked the following question at the treatment initiation visit (Day 0): 'Do you have pets living in your home?' Participants who responded 'yes' were counted.
  Participants | 26 | 10 | 36
Self-reported smoking in the participant's home [Count of Participants; unit: Participants] — Participants were asked the following question at the treatment initiation visit (Day 0): 'Does anyone smoke in your home?' Participants who responded 'yes' were counted.
  Participants | 11 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Staphylococcus Aureus Abundance on Lesional Skin, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: Staphylococcus aureus (S. aureus) abundance was measured by microbial DNA (femA qPCR) on lesional skin at Day 28, measurement is expressed in relative Colony Forming Units (rCFU)/cm^2).
  The abundance of S. aureus is summarized as the geometric mean ratio (and corresponding 95% confidence interval) between the dupilumab and placebo arms. The geometric mean ratio is reported from an ANCOVA model with fixed effects for clinical site, disease severity at Day 0 (as measured by EASI >21.1 [severe] or ≤21.1 [non-severe]) and S. aureus abundance at Day 0.
Time Frame: Day 28 (Post treatment initiation)
Population: Modified intent-to-treat: All participants who were randomized and have Staphylococcus aureus abundance measured at Day 0 and Day 28.
Measure: Geometric Mean (95% Confidence Interval); unit: Relative Colony Forming Unit (rCFU)/cm^2
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 45 | 26
Relative Colony Forming Unit (rCFU)/cm^2 | 86.01 [34.07 to 217.11] | 2608.4 [835.02 to 8147.99]
Statistical Analysis 1: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Test type: Superiority; p < 0.001, ANCOVA; Geometric Mean Ratio = 0.033, 95% CI 2-sided [0.008 to 0.131] — Dupilumab+Open Label Extension and Follow-Up arm is numerator and Placebo+Open Label Extension and Follow-Up arm is denominator

2. Secondary Outcome: Staphylococcus Aureus Abundance on Lesional Skin, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: Staphylococcus aureus (S. aureus) abundance was measured by microbial DNA (femA qPCR) on lesional skin at Days 0, 3, 7, 14, 21, 42, 77 and 112.
  The abundance of S. aureus is summarized as the geometric mean ratio (GMR) and corresponding 95% confidence interval between the dupilumab and placebo arms. The GMR is reported from a linear mixed model for repeated measures with fixed effects for S. aureus abundance on lesional skin at Day 0, treatment arm, clinical site, disease severity at Day 0 as measured by EASI ≥ 21.1 or < 21.1, time point of measurement (as a categorical variable), and an interaction term between treatment arm and pre-specified time point(s).
  A linear mixed model similar to the model specified above was fit for every time point measured. The model was used to estimate the GMR between treatment arms at Days 77 and 112 and the ratio within treatment arm between Day 77 and Day 42 and between Day 112 and Day 42.
Time Frame: Day 0 (Prior to treatment), 3, 7, 14, 21, 42, 77 and 112
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Relative Colony Forming Unit (rCFU)/cm^2
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 45 | 26
Relative Colony Forming Unit (rCFU)/cm^2
  Day 3 | 833.82 [411.45 to 1689.74] | 3028.88 [1256.63 to 7300.56]
  Day 7 | 337.48 [138.69 to 821.16] | 900.59 [290.95 to 2787.59]
  Day 14 | 205.06 [91.16 to 461.27] | 2690.79 [964.61 to 7505.96]
  Day 21 | 179.91 [80.71 to 401.02] | 2468.64 [916.89 to 6646.62]
  Day 42 | 177.79 [79.02 to 400.05] | 1112.55 [409.02 to 3026.14]
  Day 77 | 56.85 [20.44 to 158.08] | 150.81 [43.93 to 517.81]
  Day 112 | 42.35 [14.91 to 120.28] | 174.19 [53.18 to 570.53]
Statistical Analysis 1: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 3; Test type: Superiority; p = 0.019, Mixed Models Analysis; Geometric Mean Ratio = 0.28, 95% CI 2-sided [0.09 to 0.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 7; Test type: Superiority; p = 0.165, Mixed Models Analysis; Geometric Mean Ratio = 0.37, 95% CI 2-sided [0.09 to 1.51] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 14; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric Mean Ratio = 0.08, 95% CI 2-sided [0.02 to 0.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 21; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric Mean Ratio = 0.07, 95% CI 2-sided [0.02 to 0.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 42; Test type: Superiority; p = 0.004, Mixed Models Analysis; Geometric Mean Ratio = 0.16, 95% CI 2-sided [0.05 to 0.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 77; Test type: Superiority; p = 0.216, Mixed Models Analysis; Geometric Mean Ratio = 0.38, 95% CI 2-sided [0.08 to 1.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 112; Test type: Superiority; p = 0.071, Mixed Models Analysis; Geometric Mean Ratio = 0.24, 95% CI 2-sided [0.05 to 1.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 77 / Day 42; Test type: Superiority; p = 0.022, Mixed Models Analysis; Geometric Mean Ratio = 0.34, 95% CI 2-sided [0.13 to 0.85] — Day 77 is numerator and Day 42 is denominator
Statistical Analysis 9: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 112 / Day 42; Test type: Superiority; p = 0.015, Mixed Models Analysis; Geometric Mean Ratio = 0.25, 95% CI 2-sided [0.08 to 0.76] — Day 112 is numerator and Day 42 is denominator
Statistical Analysis 10: Comparison: Placebo+Open Label Extension and Follow-Up; Day 77 / Day 42; Test type: Superiority; p < 0.001, Mixed Models Analysis; Geometric Mean Ratio = 0.14, 95% CI 2-sided [0.04 to 0.41] — Day 77 is numerator and Day 42 is denominator
Statistical Analysis 11: Comparison: Placebo+Open Label Extension and Follow-Up; Day 112 / Day 42; Test type: Superiority; p = 0.006, Mixed Models Analysis; Geometric Mean Ratio = 0.16, 95% CI 2-sided [0.04 to 0.58] — Day 112 is numerator and Day 42 is denominator

3. Secondary Outcome: Staphylococcus Aureus Abundance on Non-lesional Skin, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: Staphylococcus aureus (S. aureus) abundance was measured by microbial DNA (femA qPCR) on non-lesional skin at Days 0, 3, 7, 14, 21, 28, 42, 77 and 112.
  The abundance of S. aureus is summarized as the geometric mean ratio (GMR) and corresponding 95% confidence interval between the dupilumab and placebo arms. The GMR is reported from a linear mixed model for repeated measures with fixed effects for S. aureus abundance on non-lesional skin at Day 0, treatment arm, clinical site, disease severity at Day 0 as measured by EASI ≥ 21.1 or < 21.1, time point of measurement (as a categorical variable), and an interaction term between treatment arm and pre-specified time point(s).
  A linear mixed model similar to the model specified above was fit for every time point measured. The model estimated the GMR between treatment arms at Days 77 and 112 and the ratio within treatment arm between Day 77 and Day 42 and between Day 112 and Day 42.
Time Frame: Day 0 (Prior to treatment), 3, 7, 14, 21, 28, 42, 77 and 112
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Relative Colony Forming Unit (rCFU)/cm^2
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 45 | 26
Relative Colony Forming Unit (rCFU)/cm^2
  Day 3 | 221.75 [99.74 to 493.01] | 277.21 [100.25 to 766.52]
  Day 7 | 143.19 [66.56 to 308.04] | 539.97 [201.61 to 1446.22]
  Day 14 | 118.15 [57.86 to 241.27] | 326.55 [132.38 to 805.48]
  Day 21 | 93.32 [44.33 to 196.46] | 128.56 [51.17 to 323.01]
  Day 28 | 61.67 [29.55 to 128.72] | 369.74 [145.96 to 936.60]
  Day 42 | 98.97 [44.01 to 222.55] | 191.30 [70.36 to 520.10]
  Day 77 | 86.91 [32.27 to 234.09] | 182.19 [57.37 to 578.60]
  Day 112 | 76.71 [27.37 to 214.99] | 146.35 [45.23 to 473.54]
Statistical Analysis 1: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 3; Test type: Superiority; p = 0.724, Mixed Models Analysis; Geometric Mean Ratio = 0.80, 95% CI 2-sided [0.23 to 2.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 7; Test type: Superiority; p = 0.033, Mixed Models Analysis; Geometric Mean Ratio = 0.27, 95% CI 2-sided [0.08 to 0.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 14; Test type: Superiority; p = 0.073, Mixed Models Analysis; Geometric Mean Ratio = 0.36, 95% CI 2-sided [0.12 to 1.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 21; Test type: Superiority; p = 0.579, Mixed Models Analysis; Geometric Mean Ratio = 0.73, 95% CI 2-sided [0.23 to 2.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 28; Test type: Superiority; p = 0.003, Mixed Models Analysis; Geometric Mean Ratio = 0.17, 95% CI 2-sided [0.05 to 0.53] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 42; Test type: Superiority; p = 0.297, Mixed Models Analysis; Geometric Mean Ratio = 0.52, 95% CI 2-sided [0.15 to 1.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 77; Test type: Superiority; p = 0.326, Mixed Models Analysis; Geometric Mean Ratio = 0.48, 95% CI 2-sided [0.11 to 2.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 112; Test type: Superiority; p = 0.401, Mixed Models Analysis; Geometric Mean Ratio = 0.52, 95% CI 2-sided [0.11 to 2.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 77 / Day 42; Test type: Superiority; p = 0.705, Mixed Models Analysis; Geometric Mean Ratio = 0.81, 95% CI 2-sided [0.28 to 2.40] — Day 77 is numerator and Day 42 is denominator
Statistical Analysis 10: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 112 / Day 42; Test type: Superiority; p = 0.538, Mixed Models Analysis; Geometric Mean Ratio = 0.72, 95% CI 2-sided [0.25 to 2.08] — Day 112 is numerator and Day 42 is denominator
Statistical Analysis 11: Comparison: Placebo+Open Label Extension and Follow-Up; Day 77 / Day 42; Test type: Superiority; p = 0.892, Mixed Models Analysis; Geometric Mean Ratio = 0.92, 95% CI 2-sided [0.25 to 3.34] — Day 77 is numerator and Day 42 is denominator
Statistical Analysis 12: Comparison: Placebo+Open Label Extension and Follow-Up; Day 112 / Day 42; Test type: Superiority; p = 0.624, Mixed Models Analysis; Geometric Mean Ratio = 0.74, 95% CI 2-sided [0.21 to 2.56] — Day 112 is numerator and Day 42 is denominator

4. Secondary Outcome: Transepidermal Water Loss (TEWL) of Non-lesional and Lesional Skin, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: TEWL assessment is a noninvasive in vivo measurement of water loss across the stratum corneum that is used to characterize skin barrier function. Basal TEWL =baseline measure (prior to tape stripping). An increase in TEWL values shows damage to the skin barrier function.
  Basal TEWL was measured on non-lesional and lesional skin. Basal TEWL is summarized as the mean difference between the dupilumab and placebo arms. The mean difference is reported from two linear mixed models for repeated measures (lesional and non-lesional) with fixed effects for treatment arm, basal TEWL at Day 0, clinical site, and disease severity at Day 0 as measured by EASI ≥ 21.1 or < 21.1 at Days 3, 7, 14, 21, 28, and 42. Two linear mixed models similar to the models specified above were fit for every time point measured. The model was used to estimate the mean difference between treatment arms at Days 77 and 112 and the ratio within treatment arm between Day 77 and Day 42 and between Day 112 and Day 42.
Time Frame: Day 0 (Prior to treatment), 3, 7, 14, 21, 28, 42, 77 and 112
Population: Modified intent-to-treat (all participants who were randomized and have Staphylococcus aureus abundance measured at Day 0 and Day 28) with evaluable basal TEWL at any post-baseline time point.
Measure: Mean (95% Confidence Interval); unit: g/m^2/hour
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 44 | 26
g/m^2/hour
  Day 3 - Lesional | 33.46 [28.52 to 38.39] | 42.99 [36.57 to 49.41]
  Day 7 - Lesional | 40.08 [33.79 to 46.37] | 41.15 [32.70 to 49.61]
  Day 14 - Lesional | 31.96 [27.19 to 36.74] | 31.49 [25.47 to 37.51]
  Day 21 - Lesional | 28.14 [23.25 to 33.02] | 34.11 [27.74 to 40.48]
  Day 28 - Lesional | 24.93 [19.97 to 29.89] | 32.03 [25.93 to 38.13]
  Day 42 - Lesional | 25.34 [20.58 to 30.10] | 33.33 [27.46 to 39.19]
  Day 77 - Lesional | 24.54 [18.94 to 30.13] | 25.58 [19.14 to 32.02]
  Day 112 - Lesional | 22.99 [16.79 to 29.18] | 22.82 [15.87 to 29.78]
  Day 3 - Non-lesional | 24.24 [20.87 to 27.60] | 23.55 [19.05 to 28.05]
  Day 7 - Non-lesional | 22.58 [19.60 to 25.57] | 20.23 [16.28 to 24.18]
  Day 14 - Non-lesional | 23.30 [19.90 to 26.71] | 23.20 [18.77 to 27.63]
  Day 21 - Non-lesional | 19.55 [16.54 to 22.57] | 22.86 [18.78 to 26.95]
  Day 28 - Non-lesional | 17.55 [15.08 to 20.03] | 19.31 [16.11 to 22.51]
  Day 42 - Non-lesional | 16.95 [14.50 to 19.40] | 19.12 [16.17 to 22.07]
  Day 77 - Non-lesional | 15.45 [12.60 to 18.29] | 17.55 [14.27 to 20.82]
  Day 112 - Non-lesional | 13.97 [11.55 to 16.39] | 15.86 [13.05 to 18.68]
Statistical Analysis 1: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 3, Lesional; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = -9.53, 95% CI 2-sided [-17.44 to -1.63] — Dupilumab+Open Label Extension and Follow-Up arm is minuend and Placebo+Open Label Extension and Follow-Up arm is subtrahend. (Minuend - subtrahend=difference.)
Statistical Analysis 2: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 7, Lesional; Test type: Superiority; p = 0.837, Mixed Models Analysis; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-11.47 to 9.32] — Dupilumab+Open Label Extension and Follow-Up arm is minuend and Placebo+Open Label Extension and Follow-Up arm is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 3: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 14, Lesional; Test type: Superiority; p = 0.900, Mixed Models Analysis; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-6.98 to 7.92] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 21, Lesional; Test type: Superiority; p = 0.130, Mixed Models Analysis; Mean Difference (Final Values) = -5.97, 95% CI 2-sided [-13.76 to 1.82] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 5: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 28, Lesional; Test type: Superiority; p = 0.069, Mixed Models Analysis; Mean Difference (Final Values) = -7.10, 95% CI 2-sided [-14.76 to 0.56] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 6: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 42, Lesional; Test type: Superiority; p = 0.032, Mixed Models Analysis; Mean Difference (Final Values) = -7.99, 95% CI 2-sided [-15.25 to -0.73] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 7: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 77, Lesional; Test type: Superiority; p = 0.803, Mixed Models Analysis; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-9.37 to 7.28] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 8: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 112, Lesional; Test type: Superiority; p = 0.972, Mixed Models Analysis; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-9.02 to 9.34] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 9: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 77 / Day 42, Lesional; Test type: Superiority; p = 0.933, Mixed Models Analysis; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-6.66 to 6.12] — Day 77 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 10: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 112 / Day 42, Lesional; Test type: Superiority; p = 0.563, Mixed Models Analysis; Mean Difference (Final Values) = -1.82, 95% CI 2-sided [-8.10 to 4.45] — Day 112 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 11: Comparison: Placebo+Open Label Extension and Follow-Up; Day 77 / Day 42, Lesional; Test type: Superiority; p = 0.075, Mixed Models Analysis; Mean Difference (Final Values) = -7.08, 95% CI 2-sided [-14.88 to 0.73] — Day 77 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 12: Comparison: Placebo+Open Label Extension and Follow-Up; Day 112 / Day 42, Lesional; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -9.84, 95% CI 2-sided [-17.19 to -2.48] — Day 112 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 13: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 3, Non-lesional; Test type: Superiority; p = 0.805, Mixed Models Analysis; Median Difference (Final Values) = 0.69, 95% CI 2-sided [-4.86 to 6.23] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 14: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 7, Non-lesional; Test type: Superiority; p = 0.329, Mixed Models Analysis; Mean Difference (Final Values) = 2.36, 95% CI 2-sided [-2.44 to 7.15] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 15: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 14, Non-lesional; Test type: Superiority; p = 0.970, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-5.39 to 5.60] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 16: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 21, Non-lesional; Test type: Superiority; p = 0.180, Mixed Models Analysis; Mean Difference (Final Values) = -3.31, 95% CI 2-sided [-8.18 to 1.56] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 17: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 28, Non-lesional; Test type: Superiority; p = 0.342, Mixed Models Analysis; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-5.45 to 1.94] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 18: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 42, Non-lesional; Test type: Superiority; p = 0.234, Mixed Models Analysis; Mean Difference (Final Values) = -2.17, 95% CI 2-sided [-5.81 to 1.47] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 19: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 77, Non-lesional; Test type: Superiority; p = 0.316, Mixed Models Analysis; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-6.27 to 2.07] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 20: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 112, Non-lesional; Test type: Superiority; p = 0.276, Mixed Models Analysis; Mean Difference (Final Values) = -1.89, 95% CI 2-sided [-5.37 to 1.59] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 21: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 77 / Day 42, Non-lesional; Test type: Superiority; p = 0.237, Mixed Models Analysis; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-4.19 to 1.06] — Day 77 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 22: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 112 / Day 42, Non-lesional; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -3.03, 95% CI 2-sided [-5.30 to -0.77] — Day 112 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 23: Comparison: Placebo+Open Label Extension and Follow-Up; Day 77 / Day 42, Non-lesional; Test type: Superiority; p = 0.770, Mixed Models Analysis; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-3.57 to 2.65] — Day 77 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 24: Comparison: Placebo+Open Label Extension and Follow-Up; Day 112 / Day 42, Non-lesional; Test type: Superiority; p = 0.117, Mixed Models Analysis; Mean Difference (Final Values) = -2.14, 95% CI 2-sided [-4.84 to 0.56] — Day 112 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)

5. Secondary Outcome: Transepidermal Water Loss (TEWL) Area Under the Curve (AUC) on Non-Lesional Skin, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: TEWL skin barrier assessment was assessed prior to tape stripping and repeated after 5, 10, and 15 tape strips. TEWL AUC was calculated using the trapezoidal rule and represents skin barrier integrity. An increase in TEWL values shows damage to the skin barrier function.
  TEWL AUC was measured on non-lesional skin at Days 0, 7, 14, 21, 28, 42, 77 and 112. The mean difference (between Groups) is reported from a linear mixed model for repeated measures with a random effect for participant and fixed effects for treatment arm, TEWL AUC at Day 0, clinical site, and disease severity at Day 0 as measured by EASI ≥ 21.1 or < 21.1 at Days 7, 14, 21, 28, and 42.
  A linear mixed model similar to the model specified above was fit for every time point measured. The model was used to estimate the mean difference between treatment arms at Days 77 and 112 and the mean difference within treatment arm between Day 77 and Day 42 and between Day 112 and Day 42.
Time Frame: Day 0 (Prior to treatment), 7, 14, 21, 28, 42, 77 and 112
Population: Modified intent-to-treat (all participants who were randomized and have Staphylococcus aureus abundance measured at Day 0 and Day 28) with evaluable TEWL AUC at any post-baseline time point.
Measure: Mean (95% Confidence Interval); unit: g/m^2/hour
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 43 | 26
g/m^2/hour
  Day 7 | 527.79 [466.25 to 589.33] | 442.74 [363.86 to 521.62]
  Day 14 | 504.80 [426.50 to 583.09] | 526.70 [424.66 to 628.74]
  Day 21 | 451.40 [385.72 to 517.07] | 533.89 [444.83 to 622.96]
  Day 28 | 390.92 [328.07 to 453.76] | 483.02 [405.23 to 560.81]
  Day 42 | 397.22 [341.24 to 453.20] | 445.98 [378.96 to 513.01]
  Day 77 | 363.15 [298.76 to 427.53] | 417.52 [344.23 to 490.81]
  Day 112 | 320.95 [266.16 to 375.74] | 343.92 [284.63 to 403.20]
Statistical Analysis 1: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 7; Test type: Superiority; p = 0.085, Mixed Models Analysis; Mean Difference (Final Values) = 85.05, 95% CI 2-sided [-12.02 to 182.12] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 2: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 14; Test type: Superiority; p = 0.733, Mixed Models Analysis; Mean Difference (Final Values) = -21.91, 95% CI 2-sided [-149.13 to 105.32] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 21; Test type: Superiority; p = 0.129, Mixed Models Analysis; Mean Difference (Final Values) = -82.50, 95% CI 2-sided [-189.60 to 24.61] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 28; Test type: Superiority; p = 0.057, Mixed Models Analysis; Mean Difference (Final Values) = -92.11, 95% CI 2-sided [-187.11 to 2.89] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 5: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 42; Test type: Superiority; p = 0.242, Mixed Models Analysis; Mean Difference (Final Values) = -48.76, 95% CI 2-sided [-131.52 to 34.00] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 6: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 77, Lesional; Test type: Superiority; p = 0.262, Mixed Models Analysis; Mean Difference (Final Values) = -54.37, 95% CI 2-sided [-150.24 to 41.49] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 7: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 112; Test type: Superiority; p = 0.546, Mixed Models Analysis; Mean Difference (Final Values) = -22.97, 95% CI 2-sided [-99.79 to 53.86] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 8: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 77 / Day 42; Test type: Superiority; p = 0.503, Mixed Models Analysis; Mean Difference (Final Values) = -21.80, 95% CI 2-sided [-86.34 to 42.75] — Day 77 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 9: Comparison: Dupilumab+Open Label Extension and Follow-Up; Day 112 / Day 42; Test type: Superiority; p = 0.034, Mixed Models Analysis; Mean Difference (Final Values) = -64.00, 95% CI 2-sided [-123.01 to -4.98] — Day 112 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 10: Comparison: Placebo+Open Label Extension and Follow-Up; Day 77 / Day 42; Test type: Superiority; p = 0.789, Mixed Models Analysis; Mean Difference (Final Values) = -10.29, 95% CI 2-sided [-86.63 to 66.04] — Day 77 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)
Statistical Analysis 11: Comparison: Placebo+Open Label Extension and Follow-Up; Day 112 / Day 42; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = -83.90, 95% CI 2-sided [-149.82 to -17.98] — Day 112 is minuend and Day 42 is subtrahend. (Minuend - subtrahend=difference)

6. Secondary Outcome: Transepidermal Water Loss (TEWL) Slope on Non-Lesional Skin, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: The skin tape strip collection was comprised of 1 set of 15 strips from non-lesional skin and was collected as part of the TEWL skin barrier assessment.
  The TEWL values measured at every 5 tape strips were used to model the TEWL slope. TEWL slope assesses skin barrier integrity. An increase in TEWL values shows damage to the skin barrier function.
  TEWL slope is summarized as the mean difference (and corresponding 95% confidence interval) between the dupilumab and placebo arms. The mean difference in slope for each Day is reported from a linear mixed model for repeated measures with a fixed effects for basal TEWL prior to tape stripping, treatment arm, clinical site, disease severity at Day 0 as measured by EASI ≥ 21.1 or < 21.1, tape strip number, and an interaction term between treatment arm and tape strip number.
Time Frame: Day 0 (Prior to treatment), 7, 14, 21, 28, 42, 77 and 112
Population: Modified intent-to-treat (all participants who were randomized and have Staphylococcus aureus abundance measured at Day 0 and Day 28) with evaluable TEWL at any post-baseline time point.
Measure: Number (95% Confidence Interval); unit: g/m^2/hour
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 43 | 26
g/m^2/hour
  Day 7 | 1.77 [1.25 to 2.29] | 1.84 [1.18 to 2.51]
  Day 14 | 1.56 [1.17 to 1.96] | 1.78 [1.28 to 2.28]
  Day 21 | 1.43 [0.95 to 1.91] | 1.98 [1.37 to 2.60]
  Day 28 | 1.38 [0.97 to 1.79] | 1.73 [1.23 to 2.23]
  Day 42 | 1.47 [0.96 to 1.97] | 1.76 [1.15 to 2.37]
  Day 77 | 1.15 [0.79 to 1.52] | 1.42 [0.99 to 1.85]
  Day 112 | 1.03 [0.70 to 1.36] | 1.30 [0.94 to 1.67]
Statistical Analysis 1: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 7; Test type: Superiority; p = 0.860, Mixed Models Analysis; Slope = -0.07, 95% CI 2-sided [-0.92 to 0.77] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 2: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 14; Test type: Superiority; p = 0.488, Mixed Models Analysis; Slope = -0.22, 95% CI 2-sided [-0.85 to 0.41] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 21; Test type: Superiority; p = 0.144, Mixed Models Analysis; Slope = -0.55, 95% CI 2-sided [-1.30 to 0.20] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 28; Test type: Superiority; p = 0.279, Mixed Models Analysis; Slope = -0.35, 95% CI 2-sided [-1.00 to 0.30] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 5: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 42; Test type: Superiority; p = 0.461, Mixed Models Analysis; Slope = -0.29, 95% CI 2-sided [-1.09 to 0.50] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 6: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 77, Lesional; Test type: Superiority; p = 0.345, Mixed Models Analysis; Slope = -0.27, 95% CI 2-sided [-0.84 to 0.30] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 7: Comparison: Dupilumab+Open Label Extension and Follow-Up vs Placebo+Open Label Extension and Follow-Up; Day 112; Test type: Superiority; p = 0.275, Mixed Models Analysis; Slope = -0.27, 95% CI 2-sided [-0.77 to 0.23] — [estimate comment as in outcome 4, analysis 2]

7. Secondary Outcome: Eczema Area and Severity Index (EASI) Score Within Each Treatment Group, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: EASI is a composite score (range: 0-72) measuring physical signs of atopic dermatitis, including area of involvement and severity. Severity components include: erythema, papulation, excoriation and lichenification [0=absent, 1=mild, 2=moderate, 3=severe] for each body region (head/neck, trunk, arms, legs). Area of involvement (%) is assessed for each body region. Area and severity of each body region is weighted based on size of region, and region scores are added for the total score. Scores ≤7 are considered mild, >7 and ≤21 are considered moderate, and >21 are considered severe.
  The mean EASI score in each treatment arm is reported from a linear mixed model for repeated measures with fixed effects for EASI at Day 0, treatment arm, clinical site, time point of measurement, and an interaction term between treatment arm and pre-specified time point(s), Additionally, a similar model was fit using all time points.
Time Frame: Day 0 (Prior to treatment), 3, 7, 14, 21, 28, 42, 77 and 112
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 45 | 26
units on a scale
  Day 3 | 26.52 [24.21 to 28.83] | 24.60 [21.73 to 27.46]
  Day 7 | 25.96 [23.56 to 28.36] | 24.92 [21.92 to 27.91]
  Day 14 | 20.36 [17.92 to 22.81] | 23.13 [20.08 to 26.19]
  Day 21 | 16.57 [13.98 to 19.16] | 22.75 [19.51 to 25.98]
  Day 28 | 15.09 [12.47 to 17.72] | 21.67 [18.36 to 24.99]
  Day 42 | 11.90 [9.10 to 14.70] | 20.40 [16.83 to 23.96]
  Day 77 | 8.84 [6.67 to 11.00] | 7.54 [4.89 to 10.19]
  Day 112 | 6.97 [5.19 to 8.76] | 5.53 [3.45 to 7.61]

8. Secondary Outcome: Investigator Global Assessment (IGA) Score Within Each Treatment Group, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: Investigator Global Assessment (IGA) score is a subjective scale measuring disease severity. Based on a 5-point scale from 0 (completely clear) to 4 (severe). Defined score of 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe.
  The mean IGA score in each treatment arm is reported from a linear mixed model for repeated measures with fixed effects for IGA at Day 0, treatment arm, clinical site, disease severity at Day 0 as measured by EASI ≥ 21.1 or < 21.1, time point of measurement, and an interaction term between treatment arm and pre-specified time point(s). Additionally, a similar model was fit using all time points.
Time Frame: Day 0 (Prior to treatment), 3, 7, 14, 21, 28, 42, 77 and 112
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 45 | 26
units on a scale
  Day 3 | 3.49 [3.34 to 3.64] | 3.28 [3.09 to 3.47]
  Day 7 | 3.32 [3.18 to 3.45] | 3.28 [3.11 to 3.45]
  Day 14 | 3.12 [2.96 to 3.28] | 3.16 [2.96 to 3.37]
  Day 21 | 2.86 [2.67 to 3.05] | 3.20 [2.96 to 3.44]
  Day 28 | 2.72 [2.52 to 2.92] | 3.28 [3.02 to 3.54]
  Day 42 | 2.58 [2.36 to 2.81] | 3.24 [2.95 to 3.53]
  Day 77 | 2.20 [1.92 to 2.48] | 2.20 [1.84 to 2.55]
  Day 112 | 1.94 [1.63 to 2.24] | 1.89 [1.51 to 2.27]

9. Secondary Outcome: SCORing Atopic Dermatitis (SCORAD) Score Within Each Treatment Group, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: SCORAD is a composite index comprising a) the amount/extent of body surface area affected, b) subjective symptom visual analog assessments of itch and sleep loss [itch: 0 (no itch) to 10 (worst itch imaginable) / sleep loss: 0 (no sleep loss) to 10 (worst imaginable sleep loss)], and c) 6 disease intensity assessments [dryness, erythema, edema/papulation, excoriation, lichenification and oozing/crusting, each graded from 0-3: 0 (none), 1 (mild), 2 (moderate) and 3 (severe). The score ranges from 0 (no AD present) to 103 (severe).
  The mean SCORAD score in each treatment arm is reported from a linear mixed model for repeated measures with fixed effects for SCORAD at Day 0, treatment arm, clinical site, disease severity at Day 0 as measured by EASI ≥ 21.1 or < 21.1, time point of measurement, and an interaction term between treatment arm and pre-specified time point(s). Additionally, a similar model was fit using all time points.
Time Frame: Day 0 (Prior to treatment), 3, 7, 14, 21, 28, 42, 77 and 112
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 45 | 26
units on a scale
  Day 3 | 56.91 [53.46 to 60.35] | 53.12 [48.78 to 57.46]
  Day 7 | 54.78 [51.70 to 57.86] | 54.96 [51.14 to 58.78]
  Day 14 | 46.55 [43.09 to 50.00] | 52.01 [47.66 to 56.73]
  Day 21 | 39.40 [35.53 to 43.28] | 51.87 [47.01 to 56.73]
  Day 28 | 36.34 [32.64 to 40.04] | 50.99 [46.33 to 55.66]
  Day 42 | 32.22 [28.38 to 36.06] | 51.02 [46.15 to 55.90]
  Day 77 | 27.63 [23.87 to 31.38] | 28.18 [23.53 to 32.83]
  Day 112 | 23.92 [20.25 to 27.59] | 25.01 [20.57 to 29.46]

10. Secondary Outcome: Pruritus Numerical Rating Scale (Pruritus NRS) Score Within Each Treatment Group, Dupilumab+Open Label Extension and Follow-Up Versus Placebo+Open Label Extension and Follow-Up
Description: Pruritus NRS scale is an assessment tool that is used to report the average intensity of a participant's pruritus (itch) during a 24-hour recall period. Participants were asked to report the average itch experienced during the past 24 hours on a scale of 0 - 10 [0= no itch; 10= worst imaginable itch]).
  The mean Pruritus NRS score in each treatment arm is reported from a linear mixed model for repeated measures with fixed effects for Pruritus NRS at Day 0, treatment arm, clinical site, disease severity at Day 0 as measured by EASI ≥ 21.1 or < 21.1, time point of measurement, and an interaction term between treatment arm and pre-specified time point(s). Additionally, a similar model was fit using all time points.
Time Frame: Day 0 (Prior to treatment), 3, 7, 14, 21, 28, 42, 77 and 112
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
Number analyzed (Participants) | 45 | 26
units on a scale
  Day 3 | 5.37 [4.73 to 6.01] | 5.64 [4.83 to 6.45]
  Day 7 | 5.46 [4.83 to 6.09] | 5.48 [4.69 to 6.28]
  Day 14 | 4.48 [3.91 to 5.05] | 5.29 [4.58 to 6.00]
  Day 21 | 4.20 [3.62 to 4.79] | 5.22 [4.50 to 5.93]
  Day 28 | 3.67 [3.07 to 4.28] | 5.14 [4.37 to 5.90]
  Day 42 | 3.40 [2.79 to 4.01] | 5.18 [4.41 to 5.94]
  Day 77 | 2.55 [2.05 to 3.05] | 1.88 [1.28 to 2.48]
  Day 112 | 2.38 [1.83 to 2.94] | 1.95 [1.27 to 2.64]

11. Other Pre Specified Outcome: EXPLORATORY: Composition of Bacterial Taxa
Description: 16S rRNA microbiome data (e.g., bacterial sequence reads) will be employed to identify changes in community composition and diversity at lesional and non-lesional skin sites prior to and throughout dupilumab or placebo treatment.
Time Frame: Day 0 (Prior to treatment), 16 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: EXPLORATORY: Abundance of Bacterial Taxa in Lesional and Non-lesional Skin
Description: The aim is to assess the effect of dupilumab on the skin transcriptome in lesional and non-lesional skin. Inclusion in this exploratory aim is restricted to non-University of Rochester Medical Center study participants only.
Time Frame: Day 0 (Prior to treatment), 16 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: EXPLORATORY: Gene Expression in the Skin Transcriptome in Non-lesional Skin
Description: The aim is to assess the effect of dupilumab on gene expression in the skin transcriptome of non-lesional skin.
Time Frame: Day 0 (Prior to treatment) and 7
Reporting Status: Not Posted

14. Other Pre Specified Outcome: EXPLORATORY: Gene Expression in the Skin Transcriptome in Lesional Skin
Description: The aim is to assess the effect of dupilumab on the gene expression in the skin transcriptome of lesional skin.
Time Frame: Day 0 (Prior to treatment), 7, and 21
Reporting Status: Not Posted

15. Other Pre Specified Outcome: EXPLORATORY: Lipid Profiles of Non-Lesional and Lesional Skin
Description: The aim is to assess the effect of dupilumab on lipids, which play a role in the skin barrier, will be extracted from the skin tape strips and measured using mass spectrometry methodology. Skin tape strip method allows characterization of components of the epidermis, dermis, and immune cells present in the skin.
Time Frame: Day 0 (Prior to treatment), 16 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: EXPLORATORY: Expression of S. Aureus Superantigens and Toxins on Lesional and Non-Lesional Skin
Description: The aim is to assess the effect of dupilumab on the expression of the bacterium Staphylococcus aureus (S. aureus) superantigens and toxins on lesional and non-lesional skin.
Time Frame: Day 0 (Prior to treatment), 16 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: EXPLORATORY: Confocal Imaging of Tight Junctions and Relationship to LCs in the Epidermis From Non-Lesional Skin
Description: The aim is to assess the effect of dupilumab on non-lesional skin barrier structure and Langerhans cells (LC) by confocal imaging. Inclusion in this exploratory aim is limited to University of Rochester Medical Center study participants.
Time Frame: Days 0 (Prior to treatment), 7 and 21
Reporting Status: Not Posted

18. Other Pre Specified Outcome: EXPLORATORY: Percent of Coagulase-Negative Staphylococci [CoNS] Isolates That Kill S. Aureus on Lesional and Non-Lesional Skin
Description: The aim is to assess the effect of dupilumab on the function of the skin microbiome (e.g., the ability of Coagulase-negative staphylococci isolates [CoNS] to kill S. aureus) in lesional and non-lesional skin.
Time Frame: Day 0 (Prior to treatment), 16 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: EXPLORATORY: Peripheral Blood Mononuclear Cells (PBMCs) Immunoprofiling
Description: The aim is to assess the effect of dupilumab on PBMC immunoprofiles.Flow cytometry analysis will be performed on PBMCs, using phenotyping panels to identify resting leukocyte populations, as well as T cell responses to antigens and myeloid responses to Toll-like receptor (TLR) ligands.
Time Frame: Days 0 (Prior to treatment), 14 and 28
Reporting Status: Not Posted

20. Other Pre Specified Outcome: EXPLORATORY: Levels of Serum Biomarkers (e.g. Th2 Biomarkers)
Description: The aim is to assess the effect of dupilumab on serum biomarkers (e.g. T helper type 2 [Th2] biomarkers).
Time Frame: Day 0 (Prior to treatment), 16 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: EXPLORATORY: Levels of Serum Anti-Drug Antibodies (ADA)
Description: The presence of anti-drug antibodies will be assessed and compared between intervention groups.
Time Frame: Day 0 (Prior to treatment), 16 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: EXPLORATORY: The Presence of Single Nucleotide Polymorphisms (SNPs)
Description: Towards discovery and replication of susceptibility loci in atopic dermatitis pathogenesis.
Time Frame: Day 0 (Prior to treatment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 182 days
Arm/Group | Dupilumab+Open Label Extension and Follow-Up | Placebo+Open Label Extension and Follow-Up
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/46 | 0/26
Other Adverse Events (participants affected / at risk) | 27/46 | 17/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab+Open Label Extension and Follow-Up (N=46) | Placebo+Open Label Extension and Follow-Up (N=26)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab+Open Label Extension and Follow-Up (N=46) | Placebo+Open Label Extension and Follow-Up (N=26)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 4 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 4 (4) | 3 (3)
Furuncle (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (7) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 4 (6)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 (16) | 7 (11)
Eczema (Skin and subcutaneous tissue disorders) | 12 (12) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)

LIMITATIONS AND CAVEATS:
One randomized participant did not meet criteria to be in the modified intent-to-treat (mITT) population because they withdrew prior to Day 28. Ten participants had 23 modified visits due to the coronavirus disease 2019 (COVID-19) pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03389893/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT03389893/SAP_002.pdf
  • Informed Consent Form (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03389893/ICF_003.pdf